CLINICAL TRIAL: NCT01258244
Title: Arizona Prehospital CPR Quality Improvement Project
Status: Completed | Type: Observational
Sponsor: Valleywise Health (Other)
Collaborators: Arizona Department of Health Services (Other Government); Guardian Medical Transport (Unknown); Mesa Fire Department (Unknown); Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010-118
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Out-of-Hospital Cardiac Arrest, OHCA
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Audiovisual feedback on CPR: EMS technicians will receive audiovisual feedback from the ZOLL device on depth, frequency, and interruptions to cardiac compressions
  Interventions: Other: Audiovisual Feedback

INTERVENTIONS:
Other: Audiovisual Feedback — EMTs will get audiovisual feedback on CPR technique during CPR

SUMMARY:
The quality of cardiopulmonary resuscitation (CPR) provided to patients with out-of-hospital cardiac arrest (OHCA) is often suboptimal. There now exist monitors/defibrillators that allow for the measurement and real time feedback of the quality of chest compressions and ventilations. In addition to giving the prehospital provider the benefit of real time CPR quality feedback via voice and visual cues, the CPR quality data acquired using these devices can be utilized as part of an on-going quality assurance/quality improvement program.

The first objective of the proposed project is to quantify the quality of chest compressions and ventilations provided in the state of Arizona to patients with OHCA and to determine whether the quality of CPR is related to patient outcome from OHCA.

A second objective of this project is to determine whether use of audiovisual feedback improves both CPR quality and patient outcome in the pre-hospital setting.

DETAILED DESCRIPTION:
Phase I: In the first phase of the project, the EMS systems will utilize the E-series units to treat all patients with OHCA. The audiovisual feedback prompts will be inactivated during this phase. The EMS providers will be instructed to follow the standard CCR protocol, as is currently the practice. Aside from the change in monitor/defibrillator equipment, the treatment of OHCA patients during this phase will be identical to the treatment that is currently performed. The quality of CPR will be measured using the accelerometer-based system. The data will be stored in the defibrillator and will be downloaded upon completion of the call. The first phase will be conducted for approximately 6 months from the time each site initiates the use of the E-series monitor/defibrillators.

Phase 2:In the second phase of the project, the EMS providers will undergo training on how to use the audiovisual feedback prompts. The providers will continue to treat patients according to the CCR protocol but will now receive audio and/or visual feedback on the quality of CPR that they are performing. The providers will select the preferred feedback method(s) - audio, visual or both. As in phase I, the CPR data will be stored in the defibrillator and will be downloaded upon completion of the call.

The total number of EMS personnel who will be trained is approximately 450. In Phase I, there were 219 OHCAs (80% from Mesa Fire Dept, and 20% from Guardian Medical Transport). So far in Phase II, there have been about 100 OHCAs.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medical Services personnel at 8 fire departments in AZ who treat patients with out of hospital cardiac arrest (OHCA)

Exclusion Criteria:

-

Ages: 24 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Emergency medical services providers in 4 different Arizona cities
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2010-12-07 (Actual); Primary Completion 2015-02-25 (Actual); Study Completion 2015-02-25 (Actual)

PRIMARY OUTCOMES:
Quality of chest compressions | Phase I - 6 months; Phase II - 20 months
  Depth of chest compressions, rate of chest compressions, and interruptions in chest compressions

SECONDARY OUTCOMES:
Survival to hospital discharge | Phase I - 6 months; Phase II - 20 months
  Did the patient survive to hospital discharge? (Yes or no--dichotomous measure)

CONTACTS AND LOCATIONS:
Overall Officials: Bentley J Bobrow, MD, Principal Investigator — Arizona Department of Health Services, Maricopa Integrated Health System
Locations (2):
- United States (2):
  - Guardian Medical Transport, Flagstaff, Arizona
  - Mesa Fire Department, Mesa, Arizona

REFERENCES:
- [Background] Bobrow BJ, Clark LL, Ewy GA, Chikani V, Sanders AB, Berg RA, Richman PB, Kern KB. Minimally interrupted cardiac resuscitation by emergency medical services for out-of-hospital cardiac arrest. JAMA. 2008 Mar 12;299(10):1158-65. doi: 10.1001/jama.299.10.1158. PMID 18334691
- [Background] Handley AJ, Handley SA. Improving CPR performance using an audible feedback system suitable for incorporation into an automated external defibrillator. Resuscitation. 2003 Apr;57(1):57-62. doi: 10.1016/s0300-9572(02)00400-8. PMID 12668300